CLINICAL TRIAL: NCT03691129
Title: The Studies of Yoga Efficacy and Bioactive Materials in the Blood of Korean Elderly
Brief Title: Yoga Efficacy and Bioactive Materials in the Blood of Korean Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wonryeon Cho (Other)
Responsible Party: Sponsor-Investigator, Wonryeon Cho, Associate Professor, Wonkwang University
Organization: Wonkwang University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: WonkwangU
Record Dates: First submitted 2018-09-23; First posted 2018-10-01 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Yoga; Healthy Elderly

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoga participant groups (Experimental): Yoga participant groups will practice elderly yoga for four months. We will collect their blood before and after their participation in the elderly yoga program. There will be two subgroups which are Advanced group and Beginner group.
  Interventions: Behavioral: Participation in the elderly yoga program
- Non-Yoga participant groups (No Intervention): Non-Yoga participant groups will not practice yoga for four months and will be used as the control. We will collect their blood before and after the elderly yoga program. There will be two subgroups which are Elderly group and Young group.

INTERVENTIONS:
Behavioral: Participation in the elderly yoga program — Yoga participant groups will practice elderly yoga for four months.
  Arms: Yoga participant groups

SUMMARY:
This study is conducted to verify the relationships between yoga efficacy and bioactive materials in the blood of Korean elderly.

DETAILED DESCRIPTION:
Glycoproteomics approach will be applied to verify the relationships between yoga efficacy and bioactive materials in the blood of Korean elderly.

ELIGIBILITY:
Inclusion Criteria:

* The elderly group participant over 60 years old.
* The young group participant over 20 to 57 years old.
* Individual who can read and understand Korean.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Participant who was diagnosed with cancer in the last five years.
* In case of participants leaving the yoga program after the primary blood collecting, they will be excluded from the secondary blood collecting.
* Individuals who are judged inappropriate for the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-03-23 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Measuring the number of glycoproteins in blood between before and after participation in an elderly yoga program for both the Advanced group and Beginner group | 4 months
  Glycoproteins in human plasma are known to be deeply associated with multiple diseases, cell differentiation, aging, and etc.
  The efficacy of elderly yoga will be assessed by identifying and comparing the number of glycoproteins in blood between before and after participation in an elderly yoga program for both the Advanced group and Beginner group.

CONTACTS AND LOCATIONS:
Overall Officials: Wonryeon Cho, PhD, Principal Investigator — Wonkwang University
Locations (1):
- Wonkwang University, Iksan, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No